CLINICAL TRIAL: NCT04927754
Title: Cartoon-assisted Visual/Auditory Distraction Usage in Paediatric Dental Care, Assessment of Resulting Effects on Patient Anxiety, Pain, and Behaviour.
Brief Title: Effect of Cartoon-assisted Visual/Auditory Distraction Method in Paediatric Dental Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul Medipol University Hospital (Other)
Responsible Party: Principal Investigator, Nilüfer Üstün, Assistant Professor, Istanbul Medipol University Hospital
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: E-10840098-604.01.01-E.60990
Record Dates: First submitted 2021-06-01; First posted 2021-06-16 (Actual); Last update posted 2023-08-03 (Actual); Status verified 2023-08

CONDITIONS: Behavior, Child
Keywords: dental anxiety; pain; behavior; dental care
MeSH Terms: conditions — Child Behavior; Pain; Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 (cartoon movie, then tell-show-do technique) (Experimental): Group 1: Dental treatment was carried out with showing cartoon movie as a visual/auditory distraction during the treatment in the second visit. The third visit did not consist any visual/auditory distractions, tell-show-do technique was used as a behavioural guidance technique.
  Interventions: Behavioral: Behavioral guidance; Other: Pain assessment; Other: Dental anxiety assessment
- Group 2 (tell-show-do technique, then cartoon movie) (Experimental): Group 2: Dental treatment was carried out using tell-show-do technique without any visual/auditory distraction in the second visit. The third visit consisted cartoon movie as a visual/auditory distraction.
  Interventions: Behavioral: Behavioral guidance; Other: Pain assessment; Other: Dental anxiety assessment

INTERVENTIONS:
Behavioral: Behavioral guidance — Conventional behavior guidance technique was used in one of the different treatment sessions with intervals of two weeks for both groups, and the cartoon-assisted distraction technique was used in the other. As a result, the effect of the cartoon-assisted distraction technique during dental treatment on behavior in pediatric patients was evaluated.
Other: Pain assessment — Conventional behavior guidance technique was used in one of the different treatment sessions with intervals of two weeks for both groups, and the cartoon-assisted distraction technique was used in the other. It was assessed the effect of the cartoon-assisted audio/visual distraction technique usage on paediatric patient's pain during dental care.
Other: Dental anxiety assessment — Conventional behavior guidance technique was used in one of the different treatment sessions with intervals of two weeks for both groups, and the cartoon-assisted distraction technique was used in the other. It was evaluated the effect of the cartoon-assisted audio/visual distraction technique usage on paediatric patient's dental anxiety during treatment sessions.

SUMMARY:
The hypothesis of this study was to reveal the positive effects of the visual/auditory distraction usage on anxiety, pain and behavioural control in paediatric patients. Therefore, the aim of this study was to assess the effect of the cartoon-assisted audio/visual distraction technique usage on paediatric patient's anxiety, pain and behaviour during dental care.

Children aged 4-9 years old who met inclusion criteria received restorative treatment in two sessions, with or without cartoon-assisted visual/auditory distraction technique. The parents were informed about the study following the initial dental examination of the patient and the written informed consents were obtained from parents of all participants included in the study. Following the initial dental examination, dental prophylaxis was performed to children. A behavioural assessment was done following a dental prophylaxis. Children who demonstrated a negative or positive attitude according to the behaviour assessment were selected. Although, children with definitely negative or definitely positive behavioural attitude were not selected. Subsequently, the patients were randomly assigned to two groups.

Group 1: Dental treatment was carried out with showing cartoon movie as a visual/auditory distraction during the treatment in the second visit (V2). The third visit (V3) did not consist any visual/auditory distractions.

Group 2: Dental treatment was carried out without any visual/auditory distraction in the V2. The V3 consisted cartoon movie as a visual/auditory distraction.

Paediatric patients were able to choose any of the 12 cartoon movies that have been approved by two paediatric dentists who carried out the study. Before each treatment session, parents were kindly requested to leave the operating room. Same treatment procedures were carried out in both groups during each visit in the following consecutive order. During each treatment session, corresponding measures were observed. Corresponding measures: (1) the child's anxiety; (2) the child's pain perception during local anaesthesia and treatment; (3) the child's cooperation and general behaviour.

The outcomes of the child's anxiety, pain perception and, cooperation and general behaviour for both two groups were evaluated by statistical analysis.

DETAILED DESCRIPTION:
The study was carried out in Istanbul Medipol University Department of Pedodontics, period between June 2022 - October 2022 following the ethics committee approval (REF: E-10840098-604.01.01-E.60990). The parents were informed about the study following the initial dental examination of the patient and the written informed consents were obtained from parents of all participants included in the study.

In this randomised crossover clinical study, the sample consisted of 72 children aged between 4-9 years old who applied for routine dental care in paediatric clinic.

Randomization

Following the initial dental examination eligible patients were selected (n=95) after 3 months of recruitment (June 2022 and August 2022). Each eligible patient was evaluated for the inclusion and exclusion criteria. Of these patients, 7 children demonstrated definitely negative behaviour at the first visit (V1) and 16 children did not show-up to their scheduled V1, thus 23 patients were excluded. A total of 72 patients were included the study. A randomization list was generated using online software (http://www.graphpad.com/quickcalcs/index.cfm), where consecutive patients enrolled on the study were randomized into 2 groups with an allocation ratio of 1:1. The random allocation sequence was generated by an independent researcher; thus, the operator and observer were blinded to the assignment of the study participants to the groups as follows:

Group 1: Dental treatment was carried out with showing cartoon movie as a visual/auditory distraction (group A) during the treatment in the second visit (V2). The third visit (V3) did not consist any visual/auditory distractions, tell-show-do (group B) technique was used as a behavioural guidance technique.

Group 2: Dental treatment was carried out using tell-show-do (group B) technique without any visual/auditory distraction in the V2. The V3 consisted cartoon movie as a visual/auditory distraction (group A).

Study Design This randomised crossover clinical study lasted five months with three months for recruitment and two months to allocate treatment arms, including a two-week washout period in between interventions. At the V1 following the initial dental examination, dental prophylaxis was performed using a slow-speed hand piece with a prophylaxis paste to children. A Frankl Behaviour Rating Score was assigned following dental prophylaxis. Children demonstrated a score 2 or 3 according to the Frankl Behaviour Rating Scale were selected [Frankl et al., 1962]. Subsequently, the patients were randomly assigned to as G1 (AB) or G2 (BA).

Paediatric patients were able to choose any of the 12 cartoon movies that have been approved by two paediatric dentists who carried out the study, checked for violence, slang language, and appeal to the 4-9 age range. The screen was attached to the dental unit; hence, the child could watch the cartoon movie clearly. While the same paediatric dentist performed all dental procedures in each session to remove the inter-operator variability, an independent, non-blinded observer recorded the data (all objective and subjective measures). Before each treatment session, the treatment stages were explained to the child using the tell-show-do technique the patient was requested to interrupt the treatment as little as possible. Parents were kindly requested to leave the operating room. Same treatment procedures were carried out in both groups during each visit in the following consecutive order. After the same topical anaesthesia application, mandibular block anaesthesia was performed, and followed by restoration treatment in lower primary molar tooth. Each visit time did not last longer than 30 minutes. The period between V2 and V3 was two weeks, which established as a washout period; the patients did not receive any intervention to let the effects of the previous intervention diminish.

Study Procedure Pre-operative pulse rate was retrieved by a pulse oximeter to evaluate the child's anxiety objectively. In addition, Venham Picture Test (VPT) was applied before the beginning and at the end of each visit to evaluate the child's subjective anxiety [Venham et al., 1981; Li and Lopez, 2005]. Eight cards, with two figures on each, represented anxious and non-anxious mood in the VPT. Cards were shown to the child in their numerical order and he/she was asked to choose the figure that felt closest to him/her at that moment. Choice of "anxious" figure was recorded as one, and "non-anxious" figure was recorded as zero, which totalled to a final score. According to the VPT, the score ranges from 0 (not anxious) to 8 (extremely anxious).

During the treatment, pulse rate was retrieved with the pulse oximeter at five-minute intervals starting from the local anaesthesia application. Moreover, the child's cooperation and general behaviour during treatment was rated by examiner using the Houpt Scale [Houpt et al., 1985].

Cooperation and general behaviour during treatment were evaluated using the Houpt Scale taking into consideration the patient's reactions, and interruption of treatment. The following treatment phases were evaluated, and an average was calculated to determine patient's general behaviour score.

Local anaesthesia application, The intraoral procedure with a high-speed rotary instrument, Matrix application, Restorative treatment (etch/adhesive application/polymerase/composite application with light-curing), Finishing. In order to evaluate pain perception during local anaesthesia, Sounds, Eyes and Motor Scale (SEM) scoring, which is a non-subjective method based on the observation of the physician, was used by the same examiner [Wright et al., 1991]. This method consists of two categories as comfortable (grade 1), and uncomfortable according to the patient's reactions. Uncomfortable responses were evaluated in three sub-categories: mild discomfort (grade 2), moderate discomfort (grade 3), and severe discomfort (grade 4).

Following the treatment, post-operative pulse rate and VPT were repeated. Moreover, at the end of the dental treatment, Wong-Baker FACES Pain Rating Scale was applied to the child to measure the self-reported pain during treatment [Wong and Baker, 1988]. Detailed explanation regarding the figures of the scale was provided to the child. Six faces ranging from happy to crying was shown to the child and the question "How much did you hurt during the treatment?" was asked. Based on the self-reported answer, the score was noted to the patient form.

Statistics Data was recorded to spreadsheets using Microsoft Excel (Microsoft Corporation. Redmond. WA. USA) for further analysis. NCSS (Number Cruncher Statistical System) 2007 (Kaysville, Utah, USA) software was used for statistical analysis. While evaluating the study data, descriptive statistical methods (Mean, Standard Deviation, Median, Frequency, Ratio, Minimum, and Maximum), as well as the distribution of the data, were evaluated with the Kolmogorov-Smirnov Test. Mann-Whitney U test was used to compare the quantitative data between two groups that did not show normal distribution, and Student's t-test was used in case of normal distribution. Paired test in comparisons of two periods with normal distribution; Wilcoxon test was used for comparisons between two periods (V2, V3) that did not show normal distribution. Significance was evaluated at the p<0.05 level. No subgroup analysis was carried out in this study.

ELIGIBILITY:
Inclusion Criteria:

* Systemically healthy patients without any previous dental treatment experience.
* Children who required restorative treatment in lower primary molars (pulpotomy, pulp capping, composite filling) under local anaesthesia.
* A score of 2 or 3 according to the Frankl Behaviour Rating Scale following the oral prophylaxis in the initial appointment.

Exclusion Criteria:

* Systemic disease and related continuous drug use.
* Mental and cognitive disorders, visual and auditory disabilities.
* Children demonstrated "definitely negative" or "definitely positive" behaviour (Frankl 1 or 4) following the oral prophylaxis in the initial appointment.

Ages: 4 Years to 9 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 72 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2022-10-31 (Actual); Study Completion 2022-10-31 (Actual)

PRIMARY OUTCOMES:
Child's anxiety assessment (objective) | Changes in pulse rate over 5-minute periods during procedure
  Pulse oximeter was used for objective outcomes of child's anxiety.
Child's anxiety assessment (subjective) | Change of the results of baseline Venham Picture Test compared to the end of treatment procedure up to 1 hour
  Venham Picture Test (VPT) was used for subjective outcomes of child's anxiety. Eight cards, with two figures on each, represented anxious and non-anxious mood in the VPT. Cards were shown to the child in their numerical order and he/she was asked to choose the figure that felt closest to him/her at that moment. Choice of "anxious" figure was recorded as one, and "non-anxious" figure was recorded as zero, which totalled to a final score. According to the VPT, the score ranges from 0 (not anxious) to 8 (extremely anxious).
Child's pain assessment (objective) | The first 3 minutes of the dental treatment, Sounds, Eyes and Motor Scale (SEM) scoring was used for objective outcomes.
  Sounds, Eyes and Motor Scale (SEM) scoring used for objective outcomes. This method consists of two categories as comfortable (grade 1), and uncomfortable according to the patient's reactions. Uncomfortable responses were evaluated in three sub-categories: mild discomfort (grade 2), moderate discomfort (grade 3), and severe discomfort (grade 4).
Child's pain assessment (subjective) | 5 minutes after the end of dental treatment, Wong-Baker FACES Pain Rating Scale was applied to the child to measure the self-reported pain perception.
  Wong-Baker FACES Pain Rating Scale was used for subjective outcomes. Detailed explanation regarding the figures of the scale was provided to the child. Six faces ranging from happy to crying was shown to the child and the question "How much did you hurt during the treatment?" was asked. Based on the self-reported answer, the score was noted to the patient form.
Child's cooperation assessment | Observation was done for Houpt Scale scoring for 30 minutes (during the whole procedure).
  The child's cooperation and general behaviour during treatment was rated by using the Houpt Scale. The Houpt Scale taking into consideration the patient's reactions, and interruption of treatment. The following treatment phases were evaluated (a-Local anaesthesia application, b-The intraoral procedure with a high-speed rotary instrument, c-Matrix application, d- Restorative treatment (etch/adhesive application/polymerase/composite application with light-curing), e-Finishing), and an average was calculated to determine patient's general behaviour score (1-5, higher scores mean worse outcome).

CONTACTS AND LOCATIONS:
Overall Officials: Nilüfer Üstün, Ph.D., Principal Investigator — Medipol University
Locations (1):
- Istanbul Medipol University, Faculty of Dentistry, Department of Pedodontics, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frankl SN, Shire FR, Fogels HR. Should the parent remain with the child in the dental operatory? Journal of Dentistry for Children. 1962;29(2):150-162.
- [Result] Venham LL, Goldstein M, Gaulin-Kremer E, Peteros K, Cohan J, Fairbanks J. Effectiveness of a distraction technique in managing young dental patients. Pediatr Dent. 1981 Mar;3(1):7-11. No abstract available. PMID 6951150
- [Result] Li HC, Lopez V. Children's Emotional Manifestation Scale: development and testing. J Clin Nurs. 2005 Feb;14(2):223-9. doi: 10.1111/j.1365-2702.2004.01031.x. PMID 15669931
- [Result] Houpt MI, Weiss NJ, Koenigsberg SR, Desjardins PJ. Comparison of chloral hydrate with and without promethazine in the sedation of young children. Pediatr Dent. 1985 Mar;7(1):41-6. No abstract available. PMID 3857559
- [Result] Wright GZ, Weinberger SJ, Marti R, Plotzke O. The effectiveness of infiltration anesthesia in the mandibular primary molar region. Pediatr Dent. 1991 Sep-Oct;13(5):278-83. PMID 1815200
- [Result] Wong DL, Baker CM. Pain in children: comparison of assessment scales. Pediatr Nurs. 1988 Jan-Feb;14(1):9-17. No abstract available. PMID 3344163
- [Derived] Ustun N, Akgol BB, Bayram M. Cartoon-assisted visual/auditory distraction usage in paediatric dental care, assessment of effects on patient anxiety, pain, and behaviour: a randomised crossover clinical trial. BMC Oral Health. 2025 Mar 24;25(1):425. doi: 10.1186/s12903-025-05770-4. PMID 40128690